CLINICAL TRIAL: NCT02362126
Title: Endoscopic Full Thickness Resection in the Lower GI Tract With the "Full Thickness Resection Device"- A Prospective Multicenter Trial
Brief Title: Endoscopic Full Thickness Resection in the Lower GI Tract With the "Full Thickness Resection Device"
Acronym: WALL-RESECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kliniken Ludwigsburg-Bietigheim gGmbH (Other)
Collaborators: Ovesco Endoscopy AG (Industry)
Responsible Party: Sponsor
Other Study IDs: WALL-RESECT
Record Dates: First submitted 2015-02-07; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Colorectal Adenomas; Submucosal Tumors
Keywords: Endoscopic full thickness resection; EFTR; FTRD; OTSC
MeSH Terms: interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing EFTR: Patients with non-lifting adenomas, adnomas at difficult anaotomic locations , T1-carcinomas or submucosal colorectal tumors
  Interventions: Device: Endoscopic full thickness resection (EFTR)

INTERVENTIONS:
Device: Endoscopic full thickness resection (EFTR) — Patients undergo EFTR using the FTRD

SUMMARY:
Observational prospective multicenter study to investigate efficacy and safety of endoscopic full thickness resection in the lower GI tract using a novel over-the-scope full thickness resection device.

DETAILED DESCRIPTION:
The FTRD ("Full Thickness Resection Device", Ovesco Endoscopy, Tübingen, Germany) is an over the scope device consisting of a transparent cap with a preloaded monofilament snare and and a 14 mm modified Over-the-scope Clip. The device is CE marked for full thickness resection in the lower GI tract.

The study was designed to investigate efficacy and safety of this device for full thickness resection of colorectal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y
* Adenoma with negtive lifting sign
* Adenoma involving or next to a diverticulum
* Adenoma involving or next to the appendical orifice
* T1 carcinoma with indication for endoscopic (re-)resection
* Subepithelial colorectal tumor with indication for resection

Exclusion Criteria:

* Lesions >3 cm
* T1 carcinomas with known high-risk features (submucosal infiltration>1000 um, invasion of lymphatic vessels, poor differentiation (G3))
* Lesions in the upper GI tract
* Patients with colorectal stenosis
* Patinets not able to undergo informed consent
* Pregnancy
* Patients with urgent indication for dual thrombocyte aggregation inhibition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colorectal lesions which are difficult or impossible to resect with conventional endoscopic methods
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Technical success | Immediate
  Successful enbloc- and macroscopically complete resection
R0-Resection | 3 days
  Histologically confirmed complete resection

SECONDARY OUTCOMES:
Histologically confirmed full thickness resection | 3 days
  Histologically confirmed full thickness resection
Procedure-associated complications | 3 months
  Procedure-associated complications such as bleeding or perforation
Procedure time | immediate
  Procedure time
Necessity of surgical treatment | 3 months
Residual or recurrent adenoma/carcinoma at endoscopic follow up | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karel Caca, MD, PhD, Study Chair — Klinikum Ludwigsburg, Department of Gastroenterology; Arthur R Schmidt, MD, Principal Investigator — Klinikum Ludwigsburg, Department of Gastroenterology
Locations (1):
- Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Schurr MO, Baur FE, Krautwald M, Fehlker M, Wehrmann M, Gottwald T, Prosst RL. Endoscopic full-thickness resection and clip defect closure in the colon with the new FTRD system: experimental study. Surg Endosc. 2015 Aug;29(8):2434-41. doi: 10.1007/s00464-014-3923-x. Epub 2014 Oct 16. PMID 25318369
- [Background] Schmidt A, Damm M, Caca K. Endoscopic full-thickness resection using a novel over-the-scope device. Gastroenterology. 2014 Oct;147(4):740-742.e2. doi: 10.1053/j.gastro.2014.07.045. Epub 2014 Jul 30. No abstract available. PMID 25083605
- [Derived] Kuellmer A, Behn J, Beyna T, Schumacher B, Meining A, Messmann H, Neuhaus H, Albers D, Birk M, Probst A, Faehndrich M, Frieling T, Goetz M, Thimme R, Caca K, Schmidt A. Endoscopic full-thickness resection and its treatment alternatives in difficult-to-treat lesions of the lower gastrointestinal tract: a cost-effectiveness analysis. BMJ Open Gastroenterol. 2020 Aug;7(1):e000449. doi: 10.1136/bmjgast-2020-000449. PMID 32816955
- [Derived] Schmidt A, Beyna T, Schumacher B, Meining A, Richter-Schrag HJ, Messmann H, Neuhaus H, Albers D, Birk M, Thimme R, Probst A, Faehndrich M, Frieling T, Goetz M, Riecken B, Caca K. Colonoscopic full-thickness resection using an over-the-scope device: a prospective multicentre study in various indications. Gut. 2018 Jul;67(7):1280-1289. doi: 10.1136/gutjnl-2016-313677. Epub 2017 Aug 10. PMID 28798042